CLINICAL TRIAL: NCT06906926
Title: Harmony TPV EMEA Post-Market Study
Brief Title: Harmony TPV EMEA PMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT23033CON005
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Severe Pulmonary Valve Regurgitation
Keywords: Harmony TPV; severe pulmonary regurgitation; pulmonary valve replacement
MeSH Terms: conditions — Pulmonary Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Subjects indicated for the Harmony transcatheter pulmonary heart valve treatment (Other): The Harmony TPV implant as per Standard of Care
  Interventions: Radiation: Certain imaging assessments can be non-Standard of Care

INTERVENTIONS:
Radiation: Certain imaging assessments can be non-Standard of Care — Pre-Implant CT, Chest X-Ray at discharge and any related assessments during the following up visit, can be non-standard of care depending on site's / countries.

SUMMARY:
The Harmony Transcatheter Pulmonary Valve (TPV) System is indicated for use in the management of pediatric and adult congenital heart disease patients with severe pulmonary regurgitation (i.e., severe pulmonary regurgitation as determined by echocardiography and/or pulmonary regurgitant fraction ≥ 30% as determined by cardiac magnetic resonance imaging) who have a native or surgically-repaired right ventricular outflow tract and are clinically indicated for pulmonary valve replacement as judged by the medical team.

DETAILED DESCRIPTION:
Prospective, non-randomized, multi-center, post-market interventional clinical study

ELIGIBILITY:
Inclusion Criteria:

1. Subject eligible to receive Harmony TPV System in conformity with Instructions for Use (IFU) and local regulations at time of study enrollment.
2. Subject or subject's parent(s)/legal guardian(s) must be willing and able to consent to participate in the study and will commit to completion of all follow-up requirements

Exclusion Criteria:

1. Obstruction of the central veins.
2. Planned concomitant branch pulmonary artery stenting at time of implant.
3. Subjects previously treated with an RV-PA conduit or previously implanted bioprosthesis.
4. A major or progressive non-cardiac disease (e.g. liver failure, renal failure, cancer) that results in a life expectancy of less than one year.
5. Planned implantation of the Harmony TPV in the left heart.
6. Echocardiographic evidence of intracardiac mass, thrombus, or vegetation.
7. Pre-existing prosthetic heart valve or prosthetic ring in any position
8. Subject is pregnant as confirmed by a positive pregnancy test before implant procedure for female subjects of childbearing potential.
9. Subjects that are vulnerable as defined in the Section 10.5 Subject Consent

Subject Consent Section excerpt:

* Vulnerable adults, defined as subjects incapable of giving consent, as assessed per Investigator's opinion and in consideration of vulnerable adult definition per ISO 14155, will not be included in this study.
* Any subject with mental incompetence (e.g. Alzheimer's, dementia, psychiatric disorders, developmental disorders, chromosomal abnormalities with associated cognitive impairment) should be assessed by the Investigator for vulnerable status. If pediatric or adult subject is deemed by the Investigator mentally incompetent as described above, the subject will not be included in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects without valve reintervention and with acceptable hemodynamic function composite at 6 months as defined by: | 6 months
  * Mean RVOT gradient as measured by continuous-wave Doppler echocardiography ≤40 mmHg AND
  * Pulmonary regurgitant fraction as measured by CMR <20%

SECONDARY OUTCOMES:
Percentage of subjects free from all-cause mortality at 6-months | 6 months
  Described by Kaplan-Meier statistics at 6-months.
Percentage of subjects free from reoperation at 6-months | 6 months
  Described by Kaplan-Meier statistics at 6-months
Percentage of subjects free from catheter reintervention at 6-months | 6 months
  Described by Kaplan-Meier statistics at 6-months.
Percentage of subjects free from TPV dysfunction at 6-months | 6 months
  Described by Kaplan-Meier statistics at 6-months.
Number and percentage of subjects with procedure success at 30-days | 30 days
Number and percentage of subjects with serious device-related adverse events at 6 months | 6 months
  Also described with Kaplan-Meier method for AEs of clinical interest.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ewert, Prof. Dr., Principal Investigator — TUM Klinikum Deutsches Herzzentrum
Locations (12):
- Rigshospitalet, Copenhagen, Denmark
- CHU de Bordeaux - Hôpital Cardiologique du Haut-Leveque, Bordeaux, France
- Germany (4):
  - Herz - und Diabeteszentrum NRW, Bad Oeynhausen
  - Charité - Universitätsmedizin Berlin, Berlin
  - Helios Health Institute Standort Leipzig, Leipzig
  - TUM University Hospital, Munich
- Mater Misericordiae University Hospital, Dublin, Ireland
- Schneider Children's Medical Center Israel, Petah Tikva, Israel
- Italy (2):
  - Policlinico di Sant'Orsola, Bologna
  - Azienda Ospedaliera di Padova, Padua
- Hospital General Universitario Gregorio Marañón, Madrid, Spain
- Skånes Universitetssjukhus Lund, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided